CLINICAL TRIAL: NCT00918905
Title: KOL-Fyn - an Explorative Study Wtih Telemedicine in COPD Patients at Home
Brief Title: Nurse Tele-Consultations With Discharged COPD Patients Reduce the Numbers of Readmissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Svendborg Hospital (Other)
Responsible Party: Hanne Madsen, MD, Ph.D, Consultant, Odense University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Telekol-1
Record Dates: First submitted 2009-06-03; First posted 2009-06-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pervasive healthcare; telecare; telemedicine; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Telemonitor (Experimental): Within 24 hours after the patient was discharged the telemedicine equipment was installed at the patient's home. The patients were included for four weeks followed by a visit to the outpatient clinic with a doctor. The patient was planned to have the equipment for approximately one week and had at least one follow-up phone call within the four weeks period. Telemonitoring video conferences could be made from 8 AM to 3 PM every day. The patient could call the telemedicine department in the same period of time (hot-line).
  Interventions: Device: Telemonitor
- Control group (No Intervention): No tele-monitor at home. The COPD patients discharged after an acute exacerbation living outside Svendborg or Faaborg-Midtfyn municipalities in the recruiting area were included in the control group and assigned to conventional care.

INTERVENTIONS:
Device: Telemonitor — Within 24 hours after the patient was discharged due to exacerbation in COPD the telemedicine equipment was installed at the patient's home. The patients were included for four weeks followed by a visit to the outpatient clinic with. The patient had the equipment for approximately one week and had at least one follow-up phone call. Televideo consultations could be made from 8 AM to 3 PM every day. The patient could call the telemedicine department in the same period.
  During the televideo consultations the nurse made clinical observations (i.e. dyspnoea, anxiety), measured saturation and lung function and informed the patients how to prevent exacerbations. The telemedicine consultation was agreed on with the patient and the telemedicine nurse from day to day.
  Other Names: telemonitoring; integrated care; telemedicine
  Arms: 1 Telemonitor

SUMMARY:
Patients with COPD are often admitted to the hospital with an exacerbation. It is the most common cause for admissions to medical wards. The patients are often readmitted. This is har great impact on health economy and is a significant factor to medical beds.

The aim of this study was to investigate the effect of telemedicine consultations between respiratory nurses at the hospital and COPD patients in their homes after a discharge from the hospital, which was caused by an exacerbation.

DETAILED DESCRIPTION:
Participants All patients admitted acutely to the medical ward for respiratory diseases at Odense University Hospital, Svendborg from the 4th of June 2007 until the 15th of Marts 2008 and from the 8th of August 2008 until the 6th of January 2009 were candidates if they had ECOPD defined as COPD with more dyspnoea, more cough and/or more sputum and a need for increased medication. The inclusion and exclusion criteria as mentioned in eligibility criteria.

The ECOPD patients included lived at Funen County, Denmark in the recruiting area of Odense University Hospital, Svendborg. In order to further characterize the patients at baseline, we retrieved data from the Funen County Patient Administrative System (FPAS) and the Odense University Pharmacoepidemiological Database (OPED). In brief, FPAS holds discharge diagnoses on all in-patient contacts in Funen County since 1973 and out-patient secondary care contacts since 1989. Diagnoses are coded according to the ICD8 until 1993 and ICD10 from 1994. OPED is a research database that holds information on reimbursed prescription from Funen County since 1990. All respiratory drugs are covered by the plan.

Interventions The telemedicine equipment consisted of a computer with web camera, microphone and measurement equipment with one bottom to contact to the respiratory nurse at the hospital and one alarm bottom. The nurse and the patient were able to see each other and to talk together and the nurse was able to measure saturation and perform a spirometry. The results were transferred to the hospital by a secure internet line. The equipment was especially designed to the ECOPD patients in cooperation between the OUH, Svendborg Hospital and a private company, Global IT Systems. Its popular name is "The Patient Suitcase".

Within 24 hours after the patient was discharged the telemedicine equipment was installed at the patient's home by a technician, who also collected and cleaned the equipment after use. The patients were included for four weeks followed by a visit to the outpatient clinic with a doctor. The patient was planned to have the equipment for approximately one week and had at least one follow-up phone call within the four weeks period. TVC could be made from 8 AM to 3 PM every day. The patient could call the telemedicine department in the same period of time.

During the TVC the nurse made clinical observations (i.e. dyspnoea, general condition, physical activity, anxiety), measured saturation and lung function and informed the patients how to prevent exacerbations and how to use the medication. Anxiety was estimated. The telemedicine consultation was agreed on with the patient and the telemedicine nurse from day to day. If the TVC patient were readmitted, the patient stopped with telemedicine consultations and the telemedicine equipment was collected.

All ECOPD patients who fulfilled the inclusion criteria and none of the exclusion criteria were consecutively divided into two groups due to home municipality. ECOPD patients who lived in Svendborg or Faaborg-Midtfyn municipality were included in the TVC-group and ECOPD patients from other municipalities were included in the control group.

Implementation Obviously, the study was not blinded. Every day between 8-9 AM all patients admitted to the medical ward for respiratory diseases were screened by a nurse. Patients who fulfilled the inclusion criteria's and none of the exclusion criteria's gave informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation in COPD with dyspnea, cough
* Need for medical treatment
* Age above 40 years
* Above 10 pack years
* The ability to use a phone

Exclusion Criteria:

* Communication problems
* Respiratory acidosis
* No other severe medical disease as cancer, sepsis, shock, pneumonia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
readmission to hospital | 4 weeks

SECONDARY OUTCOMES:
the duration of hospital readmission | days

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Madsen, Ph.D., Principal Investigator — Medical Department, OUH Svendborg Hospital
Locations (1):
- Medical Department, OUH Svendborg Hospital, Svendborg, Denmark